CLINICAL TRIAL: NCT06049498
Title: Efficacy and Safety of Mongolian Medicine ZhenBao Pills on Limb Function Recovery After Acute Ischemic Stroke: a Randomized Double-blinded Placebo-controlled Trial.
Brief Title: Trial of Mongolian Medicine ZhenBao Pills for Upper-limb Dysfunction After Stroke
Acronym: TREASURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-DZM-202227
Record Dates: First submitted 2023-07-24; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; Mongolian Medicine ZhenBao Pills; efficacy; safety; randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mongolian Medicine ZhenBao Pills group (Experimental): Experimental group
  Interventions: Drug: Mongolian Medicine ZhenBao Pills
- Mongolian Medicine ZhenBao Pills Placebo-controlled group (Placebo Comparator): Placebo-controlled group
  Interventions: Drug: Mongolian Medicine ZhenBao Pills Placebo

INTERVENTIONS:
Drug: Mongolian Medicine ZhenBao Pills — Mongolian Medicine ZhenBao Pills, orally, 15 pills each time, twice a day.
  Arms: Mongolian Medicine ZhenBao Pills group
Drug: Mongolian Medicine ZhenBao Pills Placebo — Mongolian Medicine ZhenBao Pills placebo, orally, 15 pills each time, twice a day.
  Arms: Mongolian Medicine ZhenBao Pills Placebo-controlled group

SUMMARY:
The trial was designed to test the hypothesis that treatment with Mongolian Medicine ZhenBao Pills has a positive effect on upper-limb motor recovery after acute ischemic stroke.

DETAILED DESCRIPTION:
The study is a randomized, double-blinded, placebo-controlled, multi-center trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (male or female ≥18 years).
2. The diagnosis of ischemic stroke should be met and the onset should be within 30 days.
3. Patients with prestroke modified Rankin scale score 0-1.
4. FAM-UE score of 20-57 at randomization.
5. The patients and legal guardians signed informed consent.

Exclusion Criteria:

1. Cranial CT or MRI findings of hemorrhage or other pathologic brain disorders, such as vascular malformations, tumors, abscesses, encephalitis, or other common non-ischemic brain diseases (e.g., multiple sclerosis).
2. Chronic liver disease or elevated ALT, AST (greater than two times the upper limit of normal), renal insufficiency or elevated blood creatinine (greater than 1.5 times the upper limit of normal).
3. Coagulation disorders or history of systemic hemorrhage.
4. Life expectancy is less than 3 months.
5. Unable to complete the study due to mental illness, cognitive or emotional impairment.
6. Suspected or known allergy to the components of the trial medication.
7. Pregnancy, breastfeeding or potential pregnancy.
8. Treatment within the last 3 months that may affect limb function, such as botulinum toxin injections or medications to improve limb motor function, etc.
9. Within three months or currently participating in another investigational study.
10. Other patients who, in the opinion of the investigator, are not suitable for participation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) scores | 90 days after randomization
  Difference in FMA-UE scores (range =0-66, with lower scores indicating more severe limb dysfunction) between baseline and 90 days after randomization.

SECONDARY OUTCOMES:
Modified Rankin scale (mRS) scores | 90 days after randomization
  Difference in the distribution of patient mRS scores (mRS scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death.)
FMA-UE scores | 30 days after randomization
  Difference in FMA-UE scores between baseline and 30 days after randomization.
The Fugl-Meyer Assessment for Lower Extremity (FMA-LE)scores | 90 days after randomization
  Difference in FMA-LE scores (range =0-34, with lower scores indicating more severe limb dysfunction) between baseline and 90 days after randomization.
National Institutes of Health Stroke Scale (NIHSS) scores | 90 days after randomization
  Difference in NIHSS scores (range =0-42, with higher scores indicating more severe strokes) between baseline and 90 days after randomization.
The Barthel index of activity of daily living (BI) | 90 days after randomization
  Difference in BI scores between baseline and 90 days after randomization. Functional independence will be measured with BI, which was a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Visual analogue scale (VAS) scores | 90 days after randomization
  Difference in VAS scores between baseline and 90 days after randomization. The patients' pain level measured with VAS, which was a conventionally used scale measuring the degree of the pain. Score of scale ranges from 0（best）to 10 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, Principal Investigator — Dongzhimen Hospital
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China